CLINICAL TRIAL: NCT01852630
Title: A Randomized, Comparative Open Label Study of Imipenem Versus Cefepime in Spontaneous Bacterial Peritonitis and to Evaluate the Risk Factors for Treatment Failure.
Brief Title: Imipenem Versus Cefepime in Spontaneous Bacterial Peritonitis and to Evaluate the Risk Factors for Treatment Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS- SBP-01
Record Dates: First submitted 2012-12-06; First posted 2013-05-14 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-07

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Cefepime; Albumins; Imipenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cefepime + Albumin (Experimental): cefepime 1g iv 8 hourly + Albumin will be given for 2 days.
  Interventions: Drug: Imipenem + Albumin
- Imipenem + Albumin (Active Comparator): Imipenem 1g iv 8 hourly + Albumin will be given for 2 days.
  Interventions: Drug: cefepime + Albumin

INTERVENTIONS:
Drug: cefepime + Albumin — cefepime + Albumin will be given for 2 days
  Arms: Imipenem + Albumin
Drug: Imipenem + Albumin — Imipenem + Albumin will be given for 2 days.
  Arms: cefepime + Albumin

SUMMARY:
1. All consecutive patients with Cirrhosis and ascites admitted to ILBS (Institute of Liver & Biliary Sciences) will be evaluated for the presence of SBP (Spontaneous Bacterial Peritonitis) by ascitic fluid examination at admission.
2. SBP (Spontaneous Bacterial Peritonitis) will be diagnosed in the presence of absolute neutrophil count (ANC >250/mm3) with/without positive ascitic fluid culture and Patients with SBP (Spontaneous Bacterial Peritonitis) included in the study will be randomized to receive cefepime or imipenem.
3. However, other SBP (Spontaneous Bacterial Peritonitis) patients not included for randomization will be given empirical therapy with 3rd generation cephalosporin (ceftriaxone).

DETAILED DESCRIPTION:
Baseline evaluation:

Baseline clinical, laboratory and disease severity parameters will be evaluated for each study patient.

1. Etiology of cirrhosis.
2. Severity of liver disease. CTP (Child-Turcotte-Pugh) score MELD (Model for End-stage Liver Disease) score MELD (Model for End-stage Liver Disease)-Na score IMSAA score
3. Decompensations/complications of CLD (Chronic Liver Disease) UGI bleed, Hepatic encephalopathy, AKI (Acute Kidney Injury) etc.
4. Laboratory investigations:

Serum electrolytes Liver function tests Kidney function tests Pro calcitonin USG/CT abdomen Complete blood counts Coagulation parameters Ascitic fluid analysis- TLC, DLC, Protein, sugar, culture, SAAG. Chest X ray PA view HBsAg and Anti-HCV and other etiological workup as available.

ELIGIBILITY:
Inclusion Criteria:

- Cirrhotic Patients with SBP (Spontaneous Bacterial Peritonitis) having any of the following risk factors would be considered as 'Difficult to Treat SBP' and would be included -

1. Nosocomial SBP: occurence of SBP (Spontaneous Bacterial Peritonitis) after 48 hours of hospital admission, or
2. Prior ascitic fluid infection with 3rd generation cephalosporin resistant organism, or
3. No response to treatment with 3rd generation cephalosporins after 48 hours.

Exclusion Criteria:

1. Age less than 18 years.
2. Cirrhotics with SBP (Spontaneous Bacterial Peritonitis) managed as outpatients.
3. Post liver transplant, HIV patients.
4. Patients on systemic chemotherapy, immunosuppressant drugs.
5. Growth of bacteria resistant to intervention drugs in ascitic fluid culture.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is the Response to treatment in each intervention group. Response is defined as 25% reduction in ANC (Absolute Neutrophil Count) from baseline. | 2 days

SECONDARY OUTCOMES:
Survival | 15 days,1 month and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ankur Jindal, MD, Principal Investigator — Institute of Liver & Biliary Sciences (ILBS)
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Jindal A, Kumar M, Bhadoria AS, Maiwall R, Sarin SK. A randomized open label study of 'imipenem vs. cefepime' in spontaneous bacterial peritonitis. Liver Int. 2016 May;36(5):677-87. doi: 10.1111/liv.12985. Epub 2015 Nov 21. PMID 26474358